CLINICAL TRIAL: NCT03830606
Title: Phase II Study of Nab-paclitaxel Plus S-1 in First-line Treatment of Advanced Biliary Tract Adenocarcinoma
Brief Title: The Efficacy and Safety of Nab-paclitaxel Plus S-1 in First-line Treatment of Advanced Biliary Tract Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-091
Record Dates: First submitted 2017-08-16; First posted 2019-02-05 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Biliary Tract Cancer
Keywords: Nab-paclitaxel, S-1, Advanced Biliary Tract Adenocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with untreated advanced biliary tract adenocarcinoma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel Plus S-1 (Experimental): Nab-paclitaxel 120 mg/m2 (D1, D8, q3w) S-1 (40mg BID for body surface area<1.25 m2; 50mg BID for body surface area of 1.25-1.5m2; and 60mg BID for body surface area>1.5 m2; D1-14, q3w)
  Interventions: Drug: Nab-paclitaxel,S-1

INTERVENTIONS:
Drug: Nab-paclitaxel,S-1 — Nab-paclitaxel 120 mg/m2 (D1, D8, q3w) and S-1 (40mg BID for body surface area < 1.25 m2; 50mg BID for body surface area of 1.25-1.5 m2; and 60mg BID for body surface area >1.5 m2; D1-14, q3w)

SUMMARY:
Advanced biliary tract adenocarcinoma has a poor prognosis with limited therapeutic options. Nab-paclitaxel plus S-1 chemotherapy will be given to untreated patients with advanced biliary tract adenocarcinoma for the first-line treatment.

DETAILED DESCRIPTION:
Gemcitabine/Nab-paclitaxel has become a standard therapy in advanced pancreatic cancer. Given the morphologic and histologic similarities between pancreatic cancer and biliary tract adenocarcinoma, nab-Paclitaxel may be a promising regimen, and S-1 has been approved for biliary tract cancer in Japan. Untreated patients with advanced biliary tract adenocarcinoma will receive Nab-paclitaxel 120 mg/m2 (D1, D8, q3w) and S-1 (40mg BID for body surface area<1.25 m2; 50mg BID for body surface area of 1.25-1.5 m2; and 60mg BID for body surface area>1.5 m2; D1-14, q3w) as the first-line treatment. The investigators will investigate the efficacy and safety of the combination treatment, and expect to provide a more effective treatment plan for patients with advanced biliary tract cancer in China.The primary endpoint is objective response rate(ORR), and the secondary endpoints are progression-free survival(PFS), overall survival(OS) and the safety.

ELIGIBILITY:
Inclusion Criteria:

* Age, years: 18-70
* Histologically and cytologically confirmed advanced biliary tract adenocarcinoma, unresectable, measurable lesions according to RECIST criteria; ECOG score of 0-1; life expectancy ≥12 weeks;
* Untreated; more than 6 months after the last adjuvant chemotherapy (does not include taxanes and S1);
* Laboratory examination within 14 days before entering the study should meet following requirements:

ANC ≥ 1.5 x 10^9/L; PLT ≥ 100 x 10^9/L; Hb ≥ 90g/L (9g/dL); AST, ALT ≤ 2.5 x ULN (with no liver metastasis), ≤ 5 x ULN（with liver metastasis); creatinine ≤ 1.5 x ULN; TBIL ≤ 1.5 x ULN

* Both male and female subjects of potential fertility have to agree effective birth control during the entire study
* Informed consent

Exclusion Criteria:

* Concurrent other effective treatment (including radiotherapy)
* Resectable patients
* Allergy history to other drugs in the same class patients with pregnancy or lactation
* Known severe internal medical diseases
* Abnormal heart function or relevant history of myocardial infarction and severe arrhythmia
* Immunocompromised patients, such as HIV positive
* Uncontrollable mental illness
* Other conditions the researchers considered ineligible for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
objective response rate（ORR） | 6 month
  Assessed by RESIST

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 month
  Assessed by Kaplan-Meier curve，From date of randomization until date of first documented PD, date of death
overall survival time (OS) | 1 year
  Assessed by Kaplan-Meier curve，From date of randomization until date of death
safety profile: assessed by CTCAE v4.0 | 1 year
  Patients with treatment-related adverse events assessed by CTCAE v4.0 to determine the tolerability of patients with Advanced Biliary Tract Adenocarcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing, China